CLINICAL TRIAL: NCT01665326
Title: Determination of Cross-Reactive Immunological Material (CRIM) Status and Longitudinal Follow-up of Individuals With Pompe Disease
Brief Title: Determination of CRIM Status and Longitudinal Follow-up of Individuals With Pompe Disease
Status: Recruiting | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00001562
Record Dates: First submitted 2012-08-13; First posted 2012-08-15 (Estimated); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Pompe Disease
Keywords: Pompe disease; Glycogen Storage Disease Type II; Acid Maltase Deficiency; CRIM Status; Acid Alpha-Glucosidase Deficiency; Alglucosidase alfa; Myozyme; Enzyme replacement therapy; Immune Tolerance Induction; Lumizyme; Immunomodulation; Anti-drug antibodies
MeSH Terms: conditions — Glycogen Storage Disease Type II | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Infantile Pompe disease: Individuals with a confirmed diagnosis of Infantile Pompe disease
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — This is a longitudinal study focused on the emerging natural history of Infantile Pompe disease, response to ERT using alglucosidase alfa (Myozyme) and response to Immune Tolerance Induction (ITI).

SUMMARY:
This is a longitudinal natural history study of Infantile Pompe disease. The investigators will regularly collect and review medical information regarding the diagnosis of Pompe disease, response to enzyme replacement (ERT) using alglucosidase alfa (Lumizyme/Myozyme) and response to immunosuppressive therapy in cases at risk for developing or those who have developed high and sustained antibodies to ERT. To follow the long-term outcomes, we will collect medical records including but not limited to the diagnosis, clinical parameters, assessments for clinical monitoring, and laboratory values including antibody testing results.

DETAILED DESCRIPTION:
Infantile-onset Pompe disease is an inherited disorder caused by lack of or defect in the enzyme acid alpha-glucosidase (GAA). GAA enzyme deficiency causes glycogen to build up and damage cells throughout the body, especially in the heart and muscles, which is normally diagnosed within the first months of life. Current treatment for Pompe disease involves enzyme replacement therapy (ERT) using the drug alglucosidase alfa (Lumizyme/Myozyme), which provides a form of the GAA enzyme to replace the enzyme that is missing or not working properly in the patient's blood.

In this study, the investigators will learn about the patient's ability to tolerate ERT. Cross-Reactive Immunological Material (CRIM) is a measurement of natural GAA production and an important factor that affects how patients respond to ERT. Children who produce some natural GAA are classified as CRIM-positive, while children who do not produce any natural GAA are classified as CRIM-negative. Children who are CRIM-positive generally tolerate ERT well. But, children who are CRIM-negative, and some children classified as CRIM-positive, have a poor response to ERT due to complications from an immune response against the drug. Treatments are currently being developed to stop this immune response and prevent complications from ERT.

This is a longitudinal natural history study of Infantile Pompe disease. The investigators will regularly collect and review medical information regarding the diagnosis of Pompe disease, response to enzyme replacement (ERT) using alglucosidase alfa (Lumizyme/Myozyme) and response to immunosuppressive therapy in cases at risk for developing or those who have developed high and sustained antibodies to ERT.

The specific aims of this study are:

1. To correlate CRIM status determined in a blood sample or cultured skin fibroblasts with GAA gene variants that are causing your child's Pompe disease.
2. To explore the clinical treatment response and natural history of CRIM-positive and CRIM-negative Pompe disease patients with and without immune modulation.
3. To investigate the role of immune response to treatment (IgG and IgE) including immune phenotyping.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of infantile, atypical or juvenile onset Pompe disease
* Must provide a written informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study subjects will be babies/children/adults with a confirmed diagnosis of infantile-onset Pompe disease who are:
  1. seen by the clinical staff of Duke Division of Medical Genetics, or
  2. whose physician or parent contacts the Duke Division of Medical Genetics with the wish to participate in this CRIM research study.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2009-09; Primary Completion 2028-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Clinical response to enzyme replacement therapy (ERT) using alglucosidase alfa (Myozyme) | Up to 18 years
  Medical records will be tracked until the patient reaches the age of 18 years to follow clinical response to ERT. This will allow us to gain an understanding of CRIM status in relation to clinical outcomes and development for these subjects.

SECONDARY OUTCOMES:
Response to Immune Tolerance Induction (ITI) | Up to 18 years
  Medical records will be tracked until the patient reaches the age of 18 years to follow clinical response to Immune Tolerance Induction (ITI) for patients who are CRIM- or CRIM+ with high antibody titers. This will allow us to increase our understanding of the history of Pompe disease in relation to treatment interventions and the role of high antibody titers in terms of patient outcome in order to develop strategies to ameliorate the immune response and other factors that may affect response to ERT.

CONTACTS AND LOCATIONS:
Overall Officials: Priya S Kishnani, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Result] Banugaria SG, Prater SN, Ng YK, Kobori JA, Finkel RS, Ladda RL, Chen YT, Rosenberg AS, Kishnani PS. The impact of antibodies on clinical outcomes in diseases treated with therapeutic protein: lessons learned from infantile Pompe disease. Genet Med. 2011 Aug;13(8):729-36. doi: 10.1097/GIM.0b013e3182174703. PMID 21637107
- [Result] Messinger YH, Mendelsohn NJ, Rhead W, Dimmock D, Hershkovitz E, Champion M, Jones SA, Olson R, White A, Wells C, Bali D, Case LE, Young SP, Rosenberg AS, Kishnani PS. Successful immune tolerance induction to enzyme replacement therapy in CRIM-negative infantile Pompe disease. Genet Med. 2012 Jan;14(1):135-42. doi: 10.1038/gim.2011.4. PMID 22237443
- [Result] Mendelsohn NJ, Messinger YH, Rosenberg AS, Kishnani PS. Elimination of antibodies to recombinant enzyme in Pompe's disease. N Engl J Med. 2009 Jan 8;360(2):194-5. doi: 10.1056/NEJMc0806809. No abstract available. PMID 19129538
- [Result] Berrier KL, Kazi ZB, Prater SN, Bali DS, Goldstein J, Stefanescu MC, Rehder CW, Botha EG, Ellaway C, Bhattacharya K, Tylki-Szymanska A, Karabul N, Rosenberg AS, Kishnani PS. CRIM-negative infantile Pompe disease: characterization of immune responses in patients treated with ERT monotherapy. Genet Med. 2015 Nov;17(11):912-8. doi: 10.1038/gim.2015.6. Epub 2015 Mar 5. PMID 25741864
- [Result] Banugaria SG, Prater SN, Patel TT, Dearmey SM, Milleson C, Sheets KB, Bali DS, Rehder CW, Raiman JA, Wang RA, Labarthe F, Charrow J, Harmatz P, Chakraborty P, Rosenberg AS, Kishnani PS. Algorithm for the early diagnosis and treatment of patients with cross reactive immunologic material-negative classic infantile pompe disease: a step towards improving the efficacy of ERT. PLoS One. 2013 Jun 25;8(6):e67052. doi: 10.1371/journal.pone.0067052. Print 2013. PMID 23825616
- [Result] Kazi ZB, Desai AK, Troxler RB, Kronn D, Packman S, Sabbadini M, Rizzo WB, Scherer K, Abdul-Rahman O, Tanpaiboon P, Nampoothiri S, Gupta N, Feigenbaum A, Niyazov DM, Sherry L, Segel R, McVie-Wylie A, Sung C, Joseph AM, Richards S, Kishnani PS. An immune tolerance approach using transient low-dose methotrexate in the ERT-naive setting of patients treated with a therapeutic protein: experience in infantile-onset Pompe disease. Genet Med. 2019 Apr;21(4):887-895. doi: 10.1038/s41436-018-0270-7. Epub 2018 Sep 14. PMID 30214072
- [Result] Desai AK, Walters CK, Cope HL, Kazi ZB, DeArmey SM, Kishnani PS. Enzyme replacement therapy with alglucosidase alfa in Pompe disease: Clinical experience with rate escalation. Mol Genet Metab. 2018 Feb;123(2):92-96. doi: 10.1016/j.ymgme.2017.12.435. Epub 2017 Dec 23. PMID 29289479
- [Result] McIntosh PT, Hobson-Webb LD, Kazi ZB, Prater SN, Banugaria SG, Austin S, Wang R, Enterline DS, Frush DP, Kishnani PS. Neuroimaging findings in infantile Pompe patients treated with enzyme replacement therapy. Mol Genet Metab. 2018 Feb;123(2):85-91. doi: 10.1016/j.ymgme.2017.10.005. Epub 2017 Oct 13. PMID 29050825
- [Result] Rairikar M, Kazi ZB, Desai A, Walters C, Rosenberg A, Kishnani PS. High dose IVIG successfully reduces high rhGAA IgG antibody titers in a CRIM-negative infantile Pompe disease patient. Mol Genet Metab. 2017 Sep;122(1-2):76-79. doi: 10.1016/j.ymgme.2017.05.006. Epub 2017 May 18. PMID 28648664
- [Result] Kazi ZB, Desai AK, Berrier KL, Troxler RB, Wang RY, Abdul-Rahman OA, Tanpaiboon P, Mendelsohn NJ, Herskovitz E, Kronn D, Inbar-Feigenberg M, Ward-Melver C, Polan M, Gupta P, Rosenberg AS, Kishnani PS. Sustained immune tolerance induction in enzyme replacement therapy-treated CRIM-negative patients with infantile Pompe disease. JCI Insight. 2017 Aug 17;2(16):e94328. doi: 10.1172/jci.insight.94328. eCollection 2017 Aug 17. PMID 28814660
- [Result] Spiridigliozzi GA, Keeling LA, Stefanescu M, Li C, Austin S, Kishnani PS. Cognitive and academic outcomes in long-term survivors of infantile-onset Pompe disease: A longitudinal follow-up. Mol Genet Metab. 2017 Jun;121(2):127-137. doi: 10.1016/j.ymgme.2017.04.014. Epub 2017 May 1. PMID 28495044
- [Result] Kazi ZB, Prater SN, Kobori JA, Viskochil D, Bailey C, Gera R, Stockton DW, McIntosh P, Rosenberg AS, Kishnani PS. Durable and sustained immune tolerance to ERT in Pompe disease with entrenched immune responses. JCI Insight. 2016 Jul 21;1(11):e86821. doi: 10.1172/jci.insight.86821. PMID 27493997
- [Result] Bali DS, Goldstein JL, Rehder C, Kazi ZB, Berrier KL, Dai J, Kishnani PS. Clinical Laboratory Experience of Blood CRIM Testing in Infantile Pompe Disease. Mol Genet Metab Rep. 2015 Dec 1;5:76-79. doi: 10.1016/j.ymgmr.2015.10.012. PMID 26693141
- [Result] Curelaru S, Desai AK, Fink D, Zehavi Y, Kishnani PS, Spiegel R. A favorable outcome in an infantile-onset Pompe patient with cross reactive immunological material (CRIM) negative disease with high dose enzyme replacement therapy and adjusted immunomodulation. Mol Genet Metab Rep. 2022 Jul 6;32:100893. doi: 10.1016/j.ymgmr.2022.100893. eCollection 2022 Sep. PMID 35813979
- [Result] Li C, Desai AK, Gupta P, Dempsey K, Bhambhani V, Hopkin RJ, Ficicioglu C, Tanpaiboon P, Craigen WJ, Rosenberg AS, Kishnani PS. Transforming the clinical outcome in CRIM-negative infantile Pompe disease identified via newborn screening: the benefits of early treatment with enzyme replacement therapy and immune tolerance induction. Genet Med. 2021 May;23(5):845-855. doi: 10.1038/s41436-020-01080-y. Epub 2021 Jan 25. PMID 33495531
- [Result] Desai AK, Baloh CH, Sleasman JW, Rosenberg AS, Kishnani PS. Benefits of Prophylactic Short-Course Immune Tolerance Induction in Patients With Infantile Pompe Disease: Demonstration of Long-Term Safety and Efficacy in an Expanded Cohort. Front Immunol. 2020 Aug 6;11:1727. doi: 10.3389/fimmu.2020.01727. eCollection 2020. PMID 32849613
- [Derived] Buckley AF, Desai AK, Ha CI, Petersen MA, Estrada JC, Water fi eld JR, Bossen EH, Kishnani PS. Outside the fiber: Endomysial stromal and capillary pathology in skeletal muscle may impede infusion therapy in infantile-onset Pompe disease. J Neuropathol Exp Neurol. 2023 Mar 20;82(4):345-362. doi: 10.1093/jnen/nlad012. PMID 36864705